CLINICAL TRIAL: NCT06835751
Title: Optimizing PrEP Among Women Who Use Drugs in Tanzania
Brief Title: Optimizing HIV Pre-exposure Prophylaxis (PrEP) Among Women Who Use Drugs in Tanzania
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00025580; R34DA058566 (NIH)
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: HIV; Mental Health; Substance Use (Drugs, Alcohol)
Keywords: HIV pre-exposure prophylaxis (PrEP); Mental health; substance use
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivational Interviewing for PreP (MI-PrEP) (Experimental): Participants randomized to this arm will receive MI-PrEP only will receive two 1-hour sessions with an intervention counselor. The first session will include information on PrEP and other HIV prevention and harm reduction strategies, and discussion on PrEP contemplation, importance, and confidence, and problem-solving around identified barriers to PrEP. The session will also include information on other available harm reduction strategies and services, including medications for opioid use disorder. The second session will focus on following up on any PrEP actions taken, challenges encountered, and problem-solving to address any challenges. Those ready to be linked to PrEP and/or harm reduction services will be offered an escort to a designated PrEP and/or opioid treatment clinic site or other harm reduction services.
  Interventions: Behavioral: Motivational Interviewing for PreP
- Common Elements Treatment Approach (CETA) + MI-PrEP (Experimental): Participants randomized to this arm will receive CETA+MI-PrEP will receive 7 to 14 weekly one-hour sessions from an intervention counselor. Similar to the MI-PrEP group, women in this study arm will receive the two 1-hour MI-PrEP sessions with an intervention counselor with linkages to PrEP and/or harm reduction services. Women will then begin CETA sessions. The CETA intervention component is a modular and flexible approach comprised of nine elements that can be combined in various ways, including different sequences, to address clients' presenting symptoms and problem areas. CETA currently includes key engagement strategies, including MI, throughout the intervention. The intervention counselor will determine the specific intervention component sessions, sequence of sessions, and dose, or frequency of sessions, based on the primary problem area identified by the participant and intervention counselor as reported in the baseline assessment survey and initial discussions.
  Interventions: Behavioral: Common Elements Treatment Approach (CETA) + MI-PrEP
- Treatment as Usual (TAU) (No Intervention): Participants randomized to this arm will receive the treatment as usual. Participants will be offered information on PrEP, including its benefits and potential side effects, and PrEP, substance use disorder treatment, including medications for opioid use disorder, overdose prevention and management, and mental health services available, as well as optional escorted linkage to a designated PrEP and/or opioid treatment clinic site. Participants will be offered linkages to a designated PrEP and/or opioid treatment clinic site or other harm reduction services, in line with current community outreach practices.

INTERVENTIONS:
Behavioral: Motivational Interviewing for PreP — Participants will receive MI-PrEP only will receive two 1-hour sessions with an intervention counselor. The first session will include information on PrEP and other HIV prevention and harm reduction strategies, and discussion on PrEP contemplation, importance, and confidence, and problem-solving around identified barriers to PrEP. The session will also include information on other available harm reduction strategies and services, including medications for opioid use disorder. The second session will focus on following up on any PrEP actions taken, challenges encountered, and problem-solving to address any challenges. Those ready to be linked to PrEP and/or harm reduction services will be offered an escort to a designated PrEP and/or opioid treatment clinic site or other harm reduction services.
  Arms: Motivational Interviewing for PreP (MI-PrEP)
Behavioral: Common Elements Treatment Approach (CETA) + MI-PrEP — Participants will receive CETA+MI-PrEP will receive 7 to 14 weekly one-hour sessions from an intervention counselor. Similar to the MI-PrEP group, women in this study arm will receive the two 1-hour MI-PrEP sessions with an intervention counselor with linkages to PrEP and/or harm reduction services. Women will then begin CETA sessions. The CETA intervention component is a modular and flexible approach comprised of nine elements that can be combined in various ways, including different sequences, to address clients' presenting symptoms and problem areas. CETA currently includes key engagement strategies, including MI, throughout the intervention. The intervention counselor will determine the specific intervention component sessions, sequence of sessions, and dose, or frequency of sessions, based on the primary problem area identified by the participant and intervention counselor as reported in the baseline assessment survey and initial discussions.
  Arms: Common Elements Treatment Approach (CETA) + MI-PrEP

SUMMARY:
This study is testing two different approaches to help women who use drugs in Tanzania take and continue using HIV prevention medication called pre-exposure prophylaxis (PrEP). Women who use drugs face a higher risk of HIV infection, but many do not start or continue PrEP due to barriers like stigma, mental health challenges, and lack of support.

The study will enroll 200 women who use drugs in Dar es Salaam, Tanzania. These women will be randomly assigned to one of three groups:

Motivational Interviewing for PrEP (MI-PrEP) Only - Women in this group will receive two one-hour counseling sessions focused on HIV prevention, PrEP education, and problem-solving to help the women start and continue using PrEP.

Common Elements Treatment Approach (CETA) + MI-PrEP - Women in this group will receive the same MI-PrEP counseling sessions plus additional mental health counseling (up to 14 sessions) tailored to the women's individual needs, addressing issues like depression, anxiety, trauma, and substance use.

Treatment as Usual (TAU) - Women in this group will receive basic information on PrEP, mental health, and harm reduction, along with optional referrals to PrEP or drug treatment clinics.

The study will evaluate feasibility of administering MI-PrEP and CETA+MI-PrEP and how well these interventions help women start and stay on PrEP, as well as the intervention's impact on mental health and drug use. Researchers will also interview participants and counselors to understand the participants and counselors experiences with the program.

The goal is to find effective ways to support PrEP use among women who use drugs and to develop a model that could be used in similar settings to reduce HIV risk. This pilot study is approved by ethics committees in the United States and Tanzania, and results will be shared with communities, policymakers, and researchers.

DETAILED DESCRIPTION:
This study is a pilot clinical trial aiming to assess the feasibility and preliminary efficacy of two interventions designed to improve PrEP engagement among women who use drugs (WWUD) in Dar es Salaam, Tanzania. The trial will enroll 200 participants who will be randomly assigned to one of three study arms: Motivational Interviewing for PrEP (MI-PrEP) only, Common Elements Treatment Approach (CETA) + MI-PrEP, or Enhanced Treatment as Usual (TAU). The study will evaluate whether these interventions can enhance PrEP uptake and adherence, while also addressing mental health and substance use challenges common among WWUD.

WWUD in Tanzania are at a heightened risk of acquiring HIV due to intersecting vulnerabilities, including drug use, high-risk sexual behaviors, and gender-based disparities. Although PrEP is a proven HIV prevention method, uptake among this population remains low due to stigma, limited healthcare access, and co-occurring mental health conditions. To address these barriers, this pilot trial will implement and evaluate MI-PrEP, a brief intervention designed to enhance motivation for PrEP use, and CETA + MI-PrEP, a more intensive mental health intervention that combines MI-PrEP with a modular, trans-diagnostic therapy addressing depression, anxiety, trauma, and substance use.

The MI-PrEP intervention will consist of two one-hour counseling sessions providing PrEP education, motivation enhancement, and problem-solving strategies. Participants in the CETA + MI-PrEP arm will receive the same MI-PrEP sessions in addition to up to 14 weekly CETA sessions tailored to individual mental health and substance use needs. The TAU control group will receive PrEP education, mental health and substance use resources, and optional referrals to PrEP and harm reduction services. The primary outcomes of the study will be feasibility, PrEP uptake, and adherence at one and six months post-intervention. Secondary outcomes include changes in depression, anxiety, PTSD symptoms, substance use behaviors, and HIV risk behaviors.

Participants will complete baseline, one-month, and six-month follow-up assessments. Quantitative data will be collected through structured surveys, while qualitative data will be obtained from in-depth interviews with a subset of trial participants and intervention counselors. Thematic analysis will be used to assess intervention feasibility, fidelity, and perceived impact. Statistical analyses, including logistic regression and mixed-effects models, will evaluate intervention effects on PrEP uptake, adherence, and mental health outcomes.

Safety protocols will be implemented to assess and manage risks related to suicide, homicide, interpersonal violence, and overdose. Ethical approvals have been obtained from the Johns Hopkins Bloomberg School of Public Health Institutional Review Board, the Muhimbili University of Health and Allied Sciences Ethics Review Committee, and the National Institute for Medical Research in Tanzania. The study also involves a Community Advisory Board (CAB) composed of WWUD and a Study Advisory Board (SAB) including representatives from academia, civil society, government agencies as well as healthcare providers and WWUD to ensure ethical and community-informed implementation.

Findings from this pilot trial will inform scalable strategies to support PrEP uptake among WWUD and other key populations at high risk for HIV infection. The results will be disseminated through community meetings, scientific conferences, and peer-reviewed publications, contributing to improved HIV prevention programming for WWUD in Tanzania and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* 18 years or older
* Non-reactive or negative HIV test result
* Self-reported drug- or sex-related HIV risk behaviors in the past six months
* Hazardous or harmful opioid use in the past six months
* Meets criteria for at least one of the following co-occurring mental health conditions: symptoms of depression (PHQ-9 >= 9), anxiety (GAD-7 >= 10), and/or PTSD (HTQ >= 40)

Exclusion Criteria:

* Reactive or positive HIV test result
* Currently taking PrEP
* Actively suicidal, homicidal, or psychotic, and needing immediate hospitalization based on safety assessments
* Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female sex
Enrollment: 200 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible participants who enroll | At baseline
  Proportion of eligible participants who enroll (Recruitment feasibility)
Proportion of target sample size enrolled | At baseline
  Proportion of target sample size enrolled in the study - Actual number of women enrolled/Planned number of women to enroll (Recruitment feasibility)
Mean proportion of planned sessions attended | 6 months post-enrollment
  Mean attendance rate, i.e., proportion of planned sessions attended (Demand & engagement)
Proportion completing all planned sessions | 6-months post-enrollment
  Proportion completing all planned sessions (Intervention delivery feasibility)
Proportion completing follow-up survey assessment | 6 months post-enrollment
  Proportion completing 6-month follow-up survey assessment (Retention feasibility)
Proportion satisfied with the intervention | 6 months post-enrollment
  Proportion satisfied or very satisfied with the intervention
Proportion of participants who report PrEP initiation | 6 months post-enrollment
  Self-reported survey measures: 1) Have you been prescribed PrEP medications? and 2) Have you received PrEP medications within 3 months of HIV testing?

SECONDARY OUTCOMES:
Change from baseline in depressive symptoms at 6 months as assessed by the PHQ-9 | Baseline and 6 months post-enrollment
  Change from baseline in depressive symptoms at 6 months post-enrolled as assessed by the Patient Health Questionnaire-9 (PHQ-9); Scoring: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe (range of 0-27)
Change from baseline in general anxiety symptoms at 6 months as assessed by GAD-7 | Baseline and 6 months post-enrollment
  Change from baseline in general anxiety symptoms at 6 months post-enrollment as assessed by the Generalized Anxiety Disorder-7 (GAD-7); 7-item scale (GAD-7) range from 0 to 21, higher scores reflect greater symptom severity.
Change from baseline in PTSD symptoms at 6 months as assessed by HTQ | Baseline and 6 months post-enrollment
  Change from baseline in post-traumatic stress disorder (PTSD) symptoms at 6 months as assessed by the Harvard Trauma Questionnaire (HTQ); Score range 16-64. Higher scores indicate higher levels of PTSD symptoms
Change from baseline in substance use risk score at 6 months as assessed by ASSIST Global Continuum of Illicit Drug Risk Score | Baseline and 6 months post-enrollment
  Change from baseline in substance use risk score at 6 months as assessed by the Alcohol, Smoking, and Substance Involvement Screening (ASSIST) Global Continuum of Illicit Drug Risk Score. Score ranges from 0 to 308, with higher scores indicating greater risk
Change from baseline in gender-based violence score at 6 months as assessed by VAWI | Baseline and 6 months post-enrollment
  Change from baseline in gender-based violence score at 6 months as assessed by the World Health Organization (WHO) Violence Against Women Instrument (VAWI). 13 Yes/No questions. Higher score reflect higher gender based violence.

CONTACTS AND LOCATIONS:
Overall Officials: Haneefa T Saleem, PhD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
The individual participant-level data that will be shared includes de-identified interview, survey, and symptom monitoring data. These data will be stored in the National Addiction & HIV Data Archive Program (NAHDAP) digital data repository of the Inter-university Consortium for Political and Social Research (ICPSR). Public use data will be accessible to registered users who agree to the ICPSR Terms of Use, while restricted access data, which may contain potentially identifying information, will be available through a virtual data enclave system for approved researchers under a restricted data contract. The rationale for sharing these data is to enable researchers to perform additional analyses to address important scientific questions related to PrEP engagement among women who use drugs, inform HIV prevention strategies, and contribute to the development of culturally appropriate interventions.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Individual participant-level data (IPD) will be available 12 months after the end of data collection
Access Criteria: Public Use Data: All deidentified study data that are not designated as restricted use will be made available as public use data to the research community via Data Sharing for Demographic Research (DSDR). Users of the public use data must register with ICPSR and agree to the Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, and requiring immediate reporting of any disclosure of study participant identity. Data users also agree not to share or redistribute any data downloads. Restricted Access Data: Data that are determined to be potentially identifying through indirect or deductive disclosure are provided under restricted data contract to users who demonstrate a valid research need and meet conditions of use. Access to restricted study data is available via a virtual data enclave system at NAHDAP/ICPSR.

REFERENCES:
- [Derived] Saleem H, Atkins K, Skavenski S, Nonyane BA, Chitamwebwa F, Mtaita S, Mwansa D, Luswetula A, Murray LK, Likindikoki S. Integrating the Common Elements Treatment Approach and motivational interviewing to improve HIV pre-exposure prophylaxis engagement among women who use drugs in Tanzania: protocol for a pilot randomised controlled trial. BMJ Open. 2026 Jan 8;16(1):e114522. doi: 10.1136/bmjopen-2025-114522. PMID 41506761